CLINICAL TRIAL: NCT04030767
Title: Evaluating Lip Repositioning for the Treatment of Excess Gingival Display With and Without Pretreatment With Botox: a Randomized Clinical Trial
Brief Title: Evaluating Lip Repositioning for the Treatment of Excess Gingival Display With and Without Pretreatment With Botox
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ola mostafa ghoniem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2261986
Record Dates: First submitted 2019-07-18; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Gingival Overgrowth
MeSH Terms: conditions — Gingival Overgrowth | interventions — incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial: Parallel group, two arm, non-inferiority trial with 1:1 allocation ratio.
Who Masked: Investigator
Masking Description: Single blinded:
  Blinding of the participants is not applicable. Blinding of the operator is not applicable. Outcome assessor (primary and secondary outcomes) & biostatistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lip repositioning technique with Botox injection. (Experimental): Botulinum toxin produces partial chemical denervation of the muscle resulting in localized reduction in muscle activity (Binder et al., 1998).
  Therefore, the technique is a useful adjunct in the esthetic improvement of the smile and provides better results when combined with resective gingival surgery(Pedron & Mangano, 2018).
  Interventions: Drug: Botox Injectable Product
- lip repositioning technique. (Active Comparator): Lip repositioning aims to limit the retraction of elevator smile muscles. Lip repositioning results in a shallow vestibuler restricting of the muscle pull; Thereby limiting the gingival display during smiling.(Makkiah, 2017) It is a less invasive, viable substitute for patients, has fewer post-operative complications and provides a faster recovery compared to orthognathic surgery(Grover, Gupta, & Luthra, 2014).
  Interventions: Drug: Botox Injectable Product

INTERVENTIONS:
Drug: Botox Injectable Product — Botulinum toxin produces partial chemical denervation of the muscle resulting in localized reduction in muscle activity
  Other Names: Xeomin

SUMMARY:
Since the introduction of the lip repositioning procedure by a number of modifications to the technique have been introduced. All these modifications were made to prevent the main complication of lip repositioning surgeries 'relapse'. Relapse was found to occur in 8% of the cases treated .

Botox injections have been suggested as a possible treatment for cases with relapse Botox acts by blocking muscular activity, however, Botulinum toxin technique has a transitory effect (6-7 months). . By combining Botox as a pretreatment and lip repositioning surgery, Botox injections maybe a useful adjunct in improving and stabilizing the results of achieved, by paralyzing the muscles during the healing period.

There are no studies, to the investigator's knowledge, exploring the use of botox combined with lip repositioning to decrease muscle pull and therefore decrease the relapse.

DETAILED DESCRIPTION:
Normal gingival display has been defined by as the gum exposure between the inferior border of upper lip and gingival margin of anterior central incisors when smiling. An exposure of gingiva around 0-2 mm when smiling, and 2-4 mm of the maxillary incisor edges when the lips are at the rest state are considered as acceptable. While more than 2 mm of gingival exposure when a person smiles is stated by experts as an excessive gingival display, or what is known as "Gummy Smile",which is more of a descriptive term than a diagnosed condition, and affects a notable proportion of the population, especially women who are affected more than men.

Many studies have stated the main causes of excessive gingival display, presenting the most important factors which may lead to having a gummy Smile. The study of Roe described that lip length and the upper lip mobility rate are the main contributing factors. The previous research stated that the exposure of teeth and gingiva depends on the integrated effects of a number of variables (increased muscle capacity, vertical maxillary excess, greater inter-labial gap at resting position, and the amount of over-jet and over-bite). Pausch & Katsoulis mentioned that abnormal gingival and maxillary anterior teeth display may take place due to numerous anatomic or functional factors, either hereditary or inborn. A narrow upper lip, an irregular eruption of teeth, excessive protuberance or vertical maxillary growth, and hypermobility of the maxillary lip and elevator muscle are common reasons for a gummy Smile. In fact, several contributing factors are affecting individuals to have a gummy Smile. Sometimes one of them is presented, although in some cases more than only one cause can be seen. Correct diagnosis of the reason leads to a proper treatment plan.

Excessive gingival display can be managed by a variety of procedures. These procedures include surgical and non-surgical methods The underlying cause of excessive gingival display or gummy Smile has the main effect on the type of procedure that will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Gummy smile more than 3mm.
2. Adults >18 years.
3. Non-smokers.
4. Patients with healthy systemic condition
5. Normal clinical crown dimensions.
6. Good oral hygiene.

Exclusion Criteria:

1. Natural dentition upper anterior
2. Pregnant or lactating women.
3. Patients with inflamed gingiva or gingival enlargement.
4. Inflammation or infection at the site of injection.
5. Patients with allergy to botulinum toxin, lactose, and albumin.
6. Concurrent use of aminoglycoside antibiotic that enhances the action of the toxin. (Jaspers, Pijpe, & Jansma, 2011)
7. < 3 mm attached gingivae that might create difficulties in flap design, stabilization and suturing.
8. Patients using anticholinesterase or other agents interfering with neuromuscular transmission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-09-20 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
change in amount of gingival display | recorded at baseline, 3, 6 ,9 months and 1 year
  Amount of gingival display (from the inferior border of the upper lip vermillion border to the gingival margin of the central incisor) will be assessed from clinical photographs obtained during active smile, with a mm ruler in place

SECONDARY OUTCOMES:
Patient satisfaction: quesionnaire | o The level of satisfaction during the followed periods (after two weeks, after two months, after six months)
  On the first follow-up visits, each patient from both groups answered a questionnaire addressing the following aspects:
  * The overall appearance.
  * Rate the improvement of their smile according to a 5-point aesthetic scale (5 = excellent, 4 = very good, 3 good, 2 = fair, 1 = poor).
  * Their willingness to repeat the treatment.